CLINICAL TRIAL: NCT01509703
Title: Respiratory Physiology Measurements Under Transnasal High Flow Therapy in Patients With Tracheostoma After Long Term Ventilation
Brief Title: Respiratory Physiology Under High Flow Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Responsible Party: Principal Investigator, Georg Nilius, Head of the department pneumology at the Helios clinic Hagen Ambrock, Helios Klinik Ambrock
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Trachea 2.0
Record Dates: First submitted 2011-12-22; First posted 2012-01-13 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Nasal High Flow Therapy; tracheotomy stent; tracheotomy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High flow therapy (Experimental)
  Interventions: Procedure: High flow therapy

INTERVENTIONS:
Procedure: High flow therapy — Each patient is treated with nasal high flow at different flow rates (15, 30, 45L/min). The order of flow rates is randomized. Each flow rate will be used for 15 minutes. A wash out time of ten minutes is planned after each phase, during which the patient uses his his individual oxygen flow.
  Other Names: AIRVO (Fisher and Paykel)

SUMMARY:
The aim of this study is to gain knowledge about effects of high flow transnasal insufflation on various breathing parameters like intratracheal pressure conditions, CO2 elimination, breathing frequency and tidal volume.

DETAILED DESCRIPTION:
Ten patients, who are supplied with a tracheostomy stent (placeholder) for reinsertions after long term ventilation will be treated for a short time during the day with the nasal high flow system AIRVO at different flow rates (15, 30, 45L/min) to estimate possible long term implications of high flow treatment.

Respiration is measured by impedance plethysmography with a calibrated belt system (Respitrace, VIASYS). Pressure and end tidal CO2 concentration is measured inside of the placeholder.

The order of the high flow rates (15, 30, 45L/min) is randomized; each flow rate is measured for 15 minutes. A wash out time of ten minutes is planned after each phase. In this time the patient breathes his individual oxygen flow rate with attention to the oxygen saturation, which should not exceed 96%. Transcutaneous PCO2 and SpO2 is monitored with TOSCA during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients in a stable weaning phase after long term ventilation
* Patients supplied with tracheostomy stent (placeholder)
* Patients in stable respiratory situation

Exclusion Criteria:

* Incapable of giving consent
* Any other severe or acute physical illness which requires intensive medical care

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Intratracheal pressure conditions | 2 hours
  The effects of high flow transnasal insufflation on intratracheal pressure conditions is measured with the Hans Rudolph Inc. pressure amplifier and continuously recorded breath by breath.

SECONDARY OUTCOMES:
Intratracheal endtidal CO2 concentration | 2 hours
  The effects of high flow transnasal insufflation on endtidal CO2 concentration is measured with the AD Instruments gas analyser and continuously recorded breath by breath.
Breathing frequency and tidal volume | 2 hours
  The effects of high flow transnasal insufflation on breathing frequency and tidal volume is measured with the Viasys Respitrace calibrated belt system and continuously recorded breath by breath.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, MD, Principal Investigator — Helios Klinik Hagen Ambrock, Germany
Locations (1):
- Helios Klinik Hagen Ambrock, Hagen, North Rhine-Westphalia, Germany